CLINICAL TRIAL: NCT03632434
Title: Acceptability and Feasibility of Transcranial Direct Current Stimulation Therapy as a Community-based Treatment for Major Depression
Brief Title: Transcranial Direct Current Stimulation Therapy for Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East London (Other)
Collaborators: Rosetrees Trust (Other); King's College London (Other); University College, London (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Cynthia Fu, College Professor of Affective Neuroscience, University of East London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1950
Record Dates: First submitted 2018-08-08; First posted 2018-08-15 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active tDCS (Experimental): 6-week course of active tDCS treatment, consisting of 5 sessions per week for the first 3 weeks followed by 2 sessions per week for 3 weeks, for a total of 21 tDCS sessions. The duration of each session is 30 minutes.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS generates a small electric current which modulates how easy it is for active brain cells to discharge. The device is a neoprene cap worn over the head, and in the cap there are two electrodes, which are small metal discs, where the current comes from.
  Other Names: tDCS

SUMMARY:
Depression is a prevalent and debilitating disorder. The most common treatments are antidepressant medications and talking therapies. However, for many individuals, these are not their treatment of choice. Furthermore, even following a full course of treatment with an antidepressant or talking therapy, over one third of patients continue to be unwell.

The novel brain stimulation treatment, transcranial direct current stimulation (tDCS), is a potential first-line treatment for major depression. The present research question is whether tDCS can be provided as a home-based treatment for major depression for adults with major depression.

DETAILED DESCRIPTION:
The novel brain stimulation treatment, transcranial direct current stimulation (tDCS), is a potential first-line treatment for major depression. tDCS generates a small electric current which modulates how easy it is for active brain cells to discharge. The device is a neoprene cap worn over the head, and in the cap there are two electrodes, which are small metal discs, where the current comes from. tDCS does not directly stimulate brain cells to cause a seizure like electroconvulsive therapy (ECT) and it does not induce brain cells to discharge like transcranial magnetic stimulation (TMS).

Clinical studies have shown that tDCS treatment could help to improve the symptoms of depression. The main side effects have been redness, skin irritation or sensations (itching, tingling or burning) under the electrodes. Less commonly reported side effects include headache or tiredness. tDCS is a portable and safe treatment.

The studies to date have mostly looked at tDCS treatment which has been provided in a research setting. This is a problem because the treatment requires daily sessions for several weeks which could limit whether individuals would be able to go every day. As tDCS is a portable and safe treatment, it could be provided in the community.

The study research question is whether tDCS could be provided as a home-based treatment for major depression. The study will include adults with major depression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depressive disorder based on DSM-5 criteria
* minimum score of 16 on Hamilton Rating Scale for Depression (HAM-D)

Exclusion Criteria:

* history of treatment-resistant depression
* comorbid psychiatric disorder
* significant risk of suicide or self harm
* any contraindications to tDCS, including implanted electronic medical devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Fu, MD PhD, Principal Investigator — University of East London
Locations (1):
- University of East London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on request.
Supporting Information: CSR
Time Frame: Starting 6 months after publication
Access Criteria: Individual access by request

REFERENCES:
- [Background] Mutz J, Edgcumbe DR, Brunoni AR, Fu CHY. Efficacy and acceptability of non-invasive brain stimulation for the treatment of adult unipolar and bipolar depression: A systematic review and meta-analysis of randomised sham-controlled trials. Neurosci Biobehav Rev. 2018 Sep;92:291-303. doi: 10.1016/j.neubiorev.2018.05.015. Epub 2018 May 12. PMID 29763711
- [Background] Mutz J, Vipulananthan V, Carter B, Hurlemann R, Fu CHY, Young AH. Comparative efficacy and acceptability of non-surgical brain stimulation for the acute treatment of major depressive episodes in adults: systematic review and network meta-analysis. BMJ. 2019 Mar 27;364:l1079. doi: 10.1136/bmj.l1079. PMID 30917990
- [Background] Woodham R, Rimmer RM, Mutz J, Fu CHY. Is tDCS a potential first line treatment for major depression? Int Rev Psychiatry. 2021 May;33(3):250-265. doi: 10.1080/09540261.2021.1879030. Epub 2021 Mar 11. PMID 33706656
- [Result] Woodham RD, Rimmer RM, Young AH, Fu CHY. Adjunctive home-based transcranial direct current stimulation treatment for major depression with real-time remote supervision: An open-label, single-arm feasibility study with long term outcomes. J Psychiatr Res. 2022 Sep;153:197-205. doi: 10.1016/j.jpsychires.2022.07.026. Epub 2022 Jul 8. PMID 35839661

RESULTS

PARTICIPANT FLOW:
Groups:
- tDCS: 6-week course of active tDCS treatment, consisting of 5 sessions per week for the first 3 weeks followed by 2 sessions per week for 3 weeks, for a total of 21 tDCS sessions. The duration of each session is 30 minutes.
  transcranial direct current stimulation: tDCS generates a small electric current which modulates how easy it is for active brain cells to discharge. The device is a neoprene cap worn over the head, and in the cap there are two electrodes, which are small metal discs, where the current comes from.
Period: Overall Study
Arm/Group | tDCS
Started | 26
Completed | 24
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | tDCS
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.85 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 16
  White and Black African | 2
  White and Asian | 1
  Any other White Background | 1
  Any other mixed/ Multiple ethnic background | 1
  Pakistani | 1
  Chinese | 1
  Any other Black/African/Caribbean background | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 26
Hamilton Depression Rating Scale score [Mean (Standard Deviation); unit: units on a scale] — Hamilton Depression Rating Scale is a clinician rated scale. Scores range from 0 - 52. Scores of 0-7 is considered to be within normal range. Entry requirement for this study was a score of 16 or greater. Higher scores indicate greater depressive symptoms.
  units on a scale | 19.12 (2.12)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: As measured by a Hamilton Depression Rating Scale score that is less than or equal to 50% of the baseline Hamilton Depression Rating Scale score. Higher scores indicate greater depressive symptoms.
Time Frame: At 6 weeks following course of tDCS treatment
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS
Number analyzed (Participants) | 24
Participants | 22

ADVERSE EVENTS:
Time Frame: Participants were asked about adverse events by researchers before and after every tDCS session for 6 weeks, then at 3 and 6 month follow-up visits. A total time frame of 7.5 months.
Description: In addition to asking participants about adverse events at every tDCS session and at follow up, the tDCS adverse events questionnaire was completed weekly during the 6-week treatment period to record adverse events that participants felt were related to the tDCS. Reported adverse events are for all participants across the full 6-weeks of treatment and indicate how many participants experienced the adverse event and how many times in total each adverse event was reported.
Arm/Group | tDCS
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 26/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS (N=26)
Headache (General disorders) | 22 (43)
Skin redness (General disorders) | 24 (104) — Skin redness at electrode site
Itching (General disorders) | 17 (46) — Itching associated with tDCS treatment
Tingling (General disorders) | 22 (94) — Tingling sensation from tDCS
Burning sensation (General disorders) | 18 (76) — Burning sensation associated with tDCS
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Scalp pain (Skin and subcutaneous tissue disorders) | 8 (16)
Sleepiness (General disorders) | 18 (52)
Trouble concentrating (General disorders) | 14 (38)
Acute mood change (Psychiatric disorders) | 8 (13)
Tingling in face (General disorders) | 1 (1)
Blurry vision (Eye disorders) | 1 (2)
Altered breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Increased anxiety (Psychiatric disorders) | 1 (1)
Flash of light in vision (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the open-label design, there was no sham treatment arm and all participants received the active tDCS treatment.

Real-time supervision at each session may have contributed to symptom improvement.

As the protocol was not designed to establish efficacy, the findings should be considered as preliminary, and a placebo sham treatment control group is required to investigate efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT03632434/Prot_SAP_000.pdf